CLINICAL TRIAL: NCT00466284
Title: Phase II Trial of Tarceva Following Concurrent Chemo-Radiotherapy as First Line Therapy in Patients With Unresectable Non-Small Cell Lung Cancer
Brief Title: Phase II Trial of Tarceva in Patients With Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Grupo Gallego de Cancer de Pulmon (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GGCP023/05-ML19497
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2007-04-27 (Estimated); Status verified 2007-04

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Tarceva (erlotinib)

SUMMARY:
A open label non- randomized Phase II trial. It is anticipated that approximately 46 patients will be treated.

STUDY OBJECTIVES

Primary: Objective response rate

Secondary: Progression free survival, Overall survival and Safety of Tarceva

DETAILED DESCRIPTION:
Study Design: Phase II trial, open label, non-randomized and multicenter.

Expected total enrollment: 46

Study start: January, 2006

Study completation: January, 2008

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years.
* Patients must have histologically confirmed diagnosis of non-small cell lung cancer, which is not surgically resectable (stage IA- IIIB).
* Measurable disease.
* Written informed consent must be obtained prior to the inclusion into the trial.
* Karnofsky performance status of 80%.
* Patients must have been treated with no prior chemotherapy or radioterapy.
* Patients must have adequate bone marrow, liver and renal function.

  * Bone Marrow: WBC > 3000 x 103/mm3,
  * Platelets > 100 x 103/mm3,
  * Hgb > 10.0 gm/dl,
  * ANC >1500 x 103/mm3,
  * Hepatic:Bilirubin < 2 mg/dl (34 µmol/l); AST, ALT, and Alkaline Phosphatase < 5 x normal,
  * Renal:Creatinine < 1.5 mg/dl (132 µmol/l).

Exclusion Criteria:

* Female patients who are pregnant or lactating.
* Patients who have used other investigational agents within 21 days prior to study entry.
* Patients who have received prior treatment with erlotinib or other anti-EGFR agent.
* Significant comorbidity.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46
Dates: Start 2006-01

PRIMARY OUTCOMES:
Objective response rate

SECONDARY OUTCOMES:
Progression free survival
Overall survival
Safety of Tarceva

CONTACTS AND LOCATIONS:
Overall Officials: Joquin Casal, MD, Principal Investigator — GGCP
Locations (1):
- Grupo Gallego de Cancer de Pulmon, Santiago de Compostela, A CORUÑA, Spain

REFERENCES:
- [Derived] Casal Rubio J, Firvida-Perez JL, Lazaro-Quintela M, Baron-Duarte FJ, Alonso-Jaudenes G, Santome L, Afonso-Afonso FJ, Amenedo M, Huidobro G, Campos-Balea B, Lopez-Vazquez MD, Vazquez S. A phase II trial of erlotinib as maintenance treatment after concurrent chemoradiotherapy in stage III non-small-cell lung cancer (NSCLC): a Galician Lung Cancer Group (GGCP) study. Cancer Chemother Pharmacol. 2014 Mar;73(3):451-7. doi: 10.1007/s00280-013-2370-z. Epub 2013 Dec 19. PMID 24352251